CLINICAL TRIAL: NCT00059098
Title: Identification of Genes Predisposing to Atherosclerosis
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1211; R01HL070150 (NIH)
Record Dates: First submitted 2003-04-17; First posted 2003-04-18 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2008-04

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases

SUMMARY:
To find genes important in the susceptibility to coronary heart disease.

DETAILED DESCRIPTION:
BACKGROUND:

Coronary heart disease (CHD) is a complex disorder constituting a major health problem in Western societies. The study assesses the unknown genetic background of CHD by investigating the most common familial dyslipidemia predisposing to CHD, familial combined hyperlipidemia (FCHL). The population prevalence of FCHL is estimated to be 1-2 percent and the disorder affects 10-20 percent of families with premature CHD. In FCHL, serum cholesterol, triglycerides, or both are elevated. Both environmental and genetic factors are suggested to affect the complex FCHL phenotype. Since the molecular basis of FCHL is unknown, a significant number of genetically predisposed individuals remain unidentified and exposed to premature CHD. The study uses samples from the genetically isolated population of Finland.

DESIGN NARRATIVE:

The investigators will use the unique study samples from the genetically isolated population of Finland and apply molecular genetic tools to first restrict the genetic locus they have identified and then to characterize the causative gene underlying the FCHL disorder on chromosome 1q21. Specifically, they first aim to further restrict the region by dissecting the different component traits. They will genotype an extended study sample consisting of all available family members of 61 FCHL families with dense sets of microsatellite markers and single nucleotide polymorphisms to fully utilize the refined quantitative phenotype information in fine mapping. Second, they aim to build a transcript map over the critical region on 1q21-q23 and to identify the causative FCHL gene among the regional candidate genes. This region on 1q21-q23 is orthologous to a region on mouse chromosome 3, where a locus (Hyplip 1) for combined hyperlipidemia has been identified. They have analyzed the human homolog of the Hyplip 1 gene but disappointingly, the human Hyplip 1 gene was found 10 Mb from the peak linkage markers and no evidence emerged for Hyplip 1 as a causative gene for FCHL. Their targets to identify the FCHL gene are currently the genes showing strongest association near the linkage peak. The FCHL gene will then be functionally characterized to prove the biological dysfunction. Characterizing one gene for FCHL would improve their understanding of molecular mechanisms of cardiovascular disease, and potentially lead to more accurate diagnosis, treatment and prevention.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-03; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leena Peltonen — University of California, Los Angeles

REFERENCES:
- [Background] Lilja HE, Suviolahti E, Soro-Paavonen A, Hiekkalinna T, Day A, Lange K, Sobel E, Taskinen MR, Peltonen L, Perola M, Pajukanta P. Locus for quantitative HDL-cholesterol on chromosome 10q in Finnish families with dyslipidemia. J Lipid Res. 2004 Oct;45(10):1876-84. doi: 10.1194/jlr.M400141-JLR200. Epub 2004 Jul 16. PMID 15258200
- [Background] Cantor RM, Chen GK, Pajukanta P, Lange K. Association testing in a linked region using large pedigrees. Am J Hum Genet. 2005 Mar;76(3):538-42. doi: 10.1086/428628. Epub 2005 Jan 18. PMID 15657872